CLINICAL TRIAL: NCT03907085
Title: The Effect of High Intensity Laser Therapy in the Management of Painful Calcaneal Spur: a Double Blind, Placebo-controlled Study
Brief Title: The Effect of High Intensity Laser Therapy in the Management of Painful Calcaneal Spur
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hilal Yeşil (Other)
Responsible Party: Sponsor-Investigator, Hilal Yeşil, Assist. Prof., Ege University
Organization: Ege University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HYHILT2019
Record Dates: First submitted 2019-04-05; First posted 2019-04-08 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Calcaneal Spur
Keywords: HILT; calcaneal spur; placebo
MeSH Terms: conditions — Heel Spur | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High intensity laser therapy (HILT) + exercise (Active Comparator): Patients received pulsed laser treatment, using a HIRO 3 device (ASA Laser, Arcugnano, Italy), five times a week for a period of three weeks, and one session per day for a total of 15 sessions. A 3-phase treatment program was performed in each session, and the patients were then given a daily exercise program once a day by a physiotherapist.
  Interventions: Other: HILT + exercise
- Placebo HILT + exercise (Placebo Comparator): Placebo therapy was applied in five sessions a week for three weeks, with a total of 15 sessions a day, with no current flowing through the device. This was followed by the exercise programs described above, performed once a day with the physiotherapist.
  Interventions: Other: Placebo HILT + exercise

INTERVENTIONS:
Other: HILT + exercise — High intensity laser therapy-Patients received pulsed laser treatment, using a HIRO 3 device (ASA Laser, Arcugnano, Italy), five times a week for a period of three weeks, and one session per day for a total of 15 sessions. A 3-phase treatment program was performed in each session, and the patients were then given a daily exercise program once a day by a physiotherapist. Exercise program; A physiotherapist-assisted exercise program was performed by the two groups, five times a week for three weeks, for approximately 25 minutes. The exercise programs consisted of stretching exercises to the plantar fascia and Achilles tendon, active range of motion (ROM) exercises, and strengthening exercises to the tibialis posterior and peroneus muscles. The patients were also taught to collect the foot and towel.
  Arms: High intensity laser therapy (HILT) + exercise
Other: Placebo HILT + exercise — Placebo HILT group; Placebo therapy was applied in five sessions a week for three weeks, with a total of 15 sessions a day, with no current flowing through the device. This was followed by the exercise programs described above, performed once a day with the physiotherapist. Exercise program; A physiotherapist-assisted exercise program was performed by the two groups, five times a week for three weeks, for approximately 25 minutes. The exercise programs consisted of stretching exercises to the plantar fascia and Achilles tendon, active range of motion (ROM) exercises, and strengthening exercises to the tibialis posterior and peroneus muscles. The patients were also taught to collect the foot and towel.
  Arms: Placebo HILT + exercise

SUMMARY:
The effect of high intensity laser therapy in the management of painful calcaneal spur: a double blind, placebo-controlled study

DETAILED DESCRIPTION:
The objective of this study was to evaluate the effect of high-intensity laser therapy (HILT) and exercise in patients with calcaneal spur. The patients were randomly assigned to receive either HILT + exercise (n=21) or placebo HILT + exercise (n=21). Pain severity (with visual analog scale (VAS) and with Roles and Maudsley score (RMS) ), functionality (with Foot and Ankle Outcome Score (FAOS)), plantar pressure measurement (with pedobarographic assesment), and quality of life (with short form-36 (SF-36)) of the patients were evaluated at baseline, at 4 weeks, and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients aged 30-75 years old with pain in the plantar region lasting for at least one month, who were sensitive to palpation and who were diagnosed with a calcaneal spur in the subcalcaneal region as shown in a lateral x-ray of the foot were included in the study.

Exclusion Criteria:

* Patients with any sign of pathology in the blood count, with an increased sedimentation rate, having undergone any physical therapy for calcaneal spur within the past six months and/or local anesthesia and/or steroid injection in the region of pain, with the presence of a pathology on the x-ray apart from calcaneal spur, pregnancy, with the presence of systemic inflammatory disease, and with a history of local trauma or a history previous HILT therapy were excluded from the study

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline visual analog scale (VAS) at 4th and 12th week. | up to 12 weeks
  The patients were asked to make an assesment of their pain between 4-12 weeks. The patients were asked to make an assessment of their pain between 0 (no pain) and 10 (severe pain).

SECONDARY OUTCOMES:
Change from baseline quality of life (short form 36 (SF-36)) at 4th and 12th weeks. | Up to12 weeks
  This is a self-administered scale, which is widely used to measure the quality of life. It was developed to measure the quality of life in patients who have physical illnesses; however, it can also be successfully used in healthy individuals and patients who have psychiatric diseases. SF-36 includes 36 items and surveys eight domains of health, such as physical functionality, physical role limitations, pain, general health, vitality, social functionality, emotional role limitations, and mental health. Total score was between 0 (no disability) and 100 (disability). Every subgroup of the questionnaire has a score scale between 0 and 100. Every increase in the subgroup of SF-36 questionnaire, which is a positive scoring system, indicates increase in quality of life related to health.
Change from baseline Foot and Ankle Outcome Score (FAOS) at 4th and 12th weeks | Up to12 weeks
  The assessment of level of functionality; was performed by Foot and Ankle Outcome Score (FAOS), which contains five subscales and which is used for the evaluation of the symptoms, pain, work-daily life, sports and recreational activities, and quality of life of patients. Each question is scored on a 5-point Likert scale (from 0 to 4), and each of the 5 subscale scores is calculated by adding the included subscale items. The raw scores are then transformed into a final score of 0 to 100 (from worst to best outcomes).
Change from baseline Roles and Maudsley Pain Score at 4th and 12th weeks. | up to 12 weeks
  General pain level assessment, performed using the Roles and Maudsley Pain Score, in which 1 point (excellent): no pain, full ROM and activity; 2 points (good): sometimes discomfort, full ROM and activity; 3 points (moderate): some pain after long-lasting activity; and 4 points (poor): activity-limiting pain.
Change from baseline static and dynamic pedobarographic evaluations at 4th and 12th weeks. | up to 12 weeks
  The plantar pressure measurement assessment was made using a pedograph (RSscan International, Olen, Belgium), and static and dynamic pedobarographic evaluations were made of all patients. For the dynamic measurement, the patient was placed on a walking platform on which the pedobarography was hidden, and was made to walk on the platform twice to obtain the normal walking speed and rhythm before measurement, and five times during the measurement. For the static measurement, the patient was placed on the pedobarograph, and the platform pressure of both feet, the upright posture of the patients, and the symmetry and parallelism of the shoulders and feet were all maintained.

CONTACTS AND LOCATIONS:
Locations (1):
- Hilal Yesil, Afyonkarahisar, Eyalet/Yerleşke, Turkey (Türkiye)